CLINICAL TRIAL: NCT05900895
Title: Phase 1b Study of Olaparib and Estradiol in Advanced ER+ Breast Cancer (PHOEBE)
Brief Title: Estradiol Plus Olaparib for Breast Cancer (PHOEBE)
Acronym: PHOEBE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mary D Chamberlin (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor-Investigator, Mary D Chamberlin, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002007
Record Dates: First submitted 2023-05-24; First posted 2023-06-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic; locally advanced; estradiol therapy; olaparib
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — olaparib; Estradiol

STUDY DESIGN:
Intervention Model Description: Single-arm, 3+3 design with a dose-expansion cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Participants receive 2 cycles of olaparib in combination with 17b-estradiol and then continue to be treated with single-agent 17b-estradiol until disease progression.
  Interventions: Drug: Olaparib; Drug: 17b-estradiol

INTERVENTIONS:
Drug: Olaparib — Participants will be treated with olaparib at the approved doses for the treatment of subtypes of breast cancer or at reduced dose/frequency for participants with moderate renal impairment.
  Other Names: Lynparza
Drug: 17b-estradiol — 17b-estradiol will be taken orally three times per day.
  Other Names: Estrace

SUMMARY:
Determine the safety and recommended Phase II dose of olaparib in combination with 17b-estradiol in post-menopausal patients with advanced ER+/HER2- breast cancer.

DETAILED DESCRIPTION:
Patients with endocrine-resistant ER+/HER2- breast cancer are eligible. Patients will be treated with the combination of 17b-estradiol and olaparib for 2 cycles, and then treated with single-agent 17b-estradiol until disease progression. Clinical benefit, progression-free survival, objective response, tumor metabolic response, and toxicity will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with ER+/HER2- breast cancer.
* Metastatic or locoregional recurrence not amenable to treatment with curative intent.
* Received ≥1 prior line of endocrine-based therapy in the advanced/metastatic setting.

Exclusion Criteria:

* During study treatment, no concurrent anti-cancer therapies are allowed with the following exceptions:

  o Anti-resorptive bone therapies (e.g., bisphosphonates, denosumab) permitted.
* Any investigational cancer therapy or systemic chemotherapy in the last 3 weeks.
* Any radiation therapy in the last 2 weeks.
* Known CNS disease, unless clinically stable for ≥ 3 months.
* Concomitant use of known strong or moderate CYP3A inhibitors.
* Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy.
* History of any of the following:

  * Deep venous thrombosis
  * Pulmonary embolism
  * Stroke
  * Acute myocardial infarction
  * Congestive heart failure
  * Previous malignancy not treated with curative intent, or with an estimated recurrence risk ≥30%
  * Severe renal impairment (creatinine clearance ≤ 30 mL/min).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Determine the Phase II dose of olaparib in combination with 17b-estradiol | 8 weeks
  Determine the safety and recommended Phase II dose of olaparib in combination with 17b-estradiol in post-menopausal patients with advanced ER+/HER2- breast cancer.

SECONDARY OUTCOMES:
Clinical benefit rate | 6 months
  The proportion of evaluable patients experiencing clinical benefit (stable disease at 24 weeks, complete or partial response per RECIST) will be measured.
Objective response rate | 6 months
  The proportion of evaluable patients experiencing objective response (complete or partial response per RECIST) will be measured.
Progression-free survival | 12 months
  Progression-free survival will be measured by measuring the length of time between the start of study treatment until the time of cancer progression or death from any cause.
Plasma Olaparib concentration | 6 hours
  The concentration of Olaparib in plasma will be measured over 6 hours.
Plasma 17b-Estradiol/Estrone concentration | 6 hours
  The concentration of 17b-Estradiol/Estrone in plasma will be measured over 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No